CLINICAL TRIAL: NCT03968588
Title: Comparative Clinical Study of Reduced Dose of Tacrolimus and Standard Dose of Mycophenolate Mofetil vs. Conventional Dose of Tacrolimus and Reduced Dose of Mycophenolate Mofetil in De Novo Renal Transplant Recipients
Brief Title: Standard- Versus Reduced-dose Tacrolimus Combined With Generic Mycophenolate Mofetil in De Novo Renal Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Chang kwon oh, Chang-Kwon Oh, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 062KTP14-1C
Record Dates: First submitted 2019-05-28; First posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Disorder Related to Renal Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reduced-dose tacrolimus + standard-dose MMF (Experimental): Tacrolimus dose was individually adjusted with a target trough blood level of between 3ng/mL and 8ng/mL throughout the study period (6 months after transplantation). MMF started within 72 hours after transplantation and the dose of MMF was 1.5~2.0g per day.
  Interventions: Drug: Tacrolimus(reduced), Mycophenolate mofetil(standard)
- standard-dose tacrolimus + reduced-dose MMF (Active Comparator): Control group, target trough blood level was between 5ng/mL and 15ng/mL throughout the study period. MMF dose was 0.5~1g per day and MMF started within 72 hours after transplantation.
  Interventions: Drug: Tacrolimus(standard), Mycophenolate mofetil(reduced)

INTERVENTIONS:
Drug: Tacrolimus(reduced), Mycophenolate mofetil(standard) — tacrolimus target trough blood level: 3~8ng/mL MMF dose: 1.5~2g/d
  Other Names: TacroBell, MY-REPT
  Arms: reduced-dose tacrolimus + standard-dose MMF
Drug: Tacrolimus(standard), Mycophenolate mofetil(reduced) — tacrolimus target trough blood level: 5~15ng/mL MMF dose: 0.5~1g/d
  Other Names: TacroBell, MY-REPT
  Arms: standard-dose tacrolimus + reduced-dose MMF

SUMMARY:
A prospective, multicenter, open-label, randomized and parallel-group clinical trial was conducted at four transplant centers in Korea. This clinical study was designed to compare the efficacy and tolerability of reduced-dose tacrolimus with standard-dose mycophenolate mofetil (MMF) versus standard-dose tacrolimus with reduced-dose MMF.

DETAILED DESCRIPTION:
A prospective, multicenter, open-label, randomized and parallel-group clinical trial was conducted at four transplant centers in Korea. The total sample size was 108 and eligible patients were randomly assigned in a 1:1 ratio to either study or control group. For six months study period, graft function, the incidence of efficacy failure and adverse events were compared.

The total sample size was 108 and eligible patients were randomly assigned in a 1:1 ratio to either study or control group: The study group (reduced-dose tacrolimus + standard-dose MMF) or the control group (standard-dose tacrolimus + reduced-dose MMF). Restricted block randomization was applied to this study and both the enrolled subjects and care providers were blinded until randomization was done. A difference in the mean estimated glomerular filtration rates (eGFR) of 16 mL/min/1.73m2 was considered a clinically meaningful margin of non-inferiority. A sample size of 108 for both groups was calculated for the primary endpoint by assuming a significance level of 0.025 with a power of at least 95% and adjusted for a potential dropout rate of 20%.

The primary efficacy endpoint was the renal graft function assessed with eGFR by MDRD formula at 6 months post-transplant. The secondary endpoints included (1) the incidence of treatment failure that included biopsy-confirmed acute rejection (BCAR), graft loss, death, or loss to follow-up until 6 months post-transplant; (2) recipients and grafts' survival rates; (3) 24-hour urine proteinuria and creatinine clearance at 6 months post-transplant. Recipients with clinical findings suggestive of acute rejection underwent biopsies before initiation or within 48 hours of anti-rejection therapy and biopsy specimens were graded according to Banff Classification criteria.

Safety endpoints included (1) all adverse event defined as any medical occurrence including worsening of a preexisting medical condition; (2) opportunistic infections; (3) malignancies; (4) abnormal laboratory findings; and (5) any abnormal physical findings or vital signs. Severe adverse events were defined as any adverse events with undesirable signs, symptoms, or medical conditions that met any one of the following criteria: 1) was fatal or life-threatening, 2) resulted in persistent or significant disability/incapacity, 3) required hospitalization or the prolongation of existing hospitalization, 4) was a congenital anomaly/birth defect, or 5) was an important medical event that might deteriorate the patient and require medical or surgical intervention to prevent one of the other outcomes listed above.18 All adverse events were coding using WHOART 2009 version.

ELIGIBILITY:
Inclusion Criteria:

* Recipients (aged 20-65) of a single (first or second) renal allograft from living or deceased donor.

Exclusion Criteria:

* comprised of recipients with multiple organ transplants
* double kidney transplant or organs donated after cardiac death
* recipients previously organ transplanted except kidney
* ABO-incompatible transplants
* recipients with antibodies against the human leukocyte antigens of the donor organ
* history of malignancy in the previous 5 years (except successfully treated localized non-melanoma skin cancer and thyroid cancer)
* leukocyte counts of less than 2,500 per μL, or neutrophils less than 1,500 per μL, or platelets less than 50,000 per μL
* evidence of active systemic infection requiring the use of antibiotics, human immunodeficiency virus infection, or chronic active hepatitis B or C

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-07-29 (Actual); Primary Completion 2016-11-11 (Actual); Study Completion 2017-06-14 (Actual)

PRIMARY OUTCOMES:
renal graft function | 6 months post-transplant
  assessed with eGFR by MDRD formula

SECONDARY OUTCOMES:
incidence of treatment failure | 6 months post-transplant
  biopsy-confirmed acute rejection (BCAR), graft loss, death, or loss
recipients and grafts' survival rates | 6 months post-transplant
  recipients and grafts' survival rates
24-hour urine proteinuria and creatinine clearance | 6 months post-transplant
  24-hour urine proteinuria and creatinine clearance

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Kwon Oh, M.D, Principal Investigator — Department of surgery, Ajou University School of Medicine
Locations (4):
- South Korea (4):
  - Chonbuk National University Hospital, Jeonju
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Ajou University Hospital, Suwon

IPD SHARING:
Plan to Share IPD: No